CLINICAL TRIAL: NCT05156944
Title: Effect of Physiotherapy in Patients Presenting to the Emergency Department After a Fall. A Brief Intervention Focusing on Patient Reported Outcomes
Brief Title: Effect of Physiotherapy in Patients Presenting to the Emergency Department After a Fall
Acronym: EPAC-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021-02165; am21Bingisser2
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Fear of Falling
Keywords: fall; Ground Level Fall" (GLF); physiotherapy intervention; short International Falls efficacy scale (sFES-I)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The study intervention is a brief physiotherapeutic assessment, a brief information on the expected course of the condition, and a brief instruction on self-management, including two exercises for daily self-guided therapy.
  Interventions: Other: physiotherapeutic intervention
- control group (No Intervention): The control group will receive written information on the expected course of the condition, written instructions on self-management and written instructions on exercises for daily self-guided therapy.

INTERVENTIONS:
Other: physiotherapeutic intervention — The intervention consists of a brief physiotherapeutic assessment, the short physical performance battery, a brief information on the expected course of the condition, a check of fall hazards at home using the "Bundesamt für Unfallverhütung" (bfu) checklist, and instructions on self-management (eg. staying active, adaptation of behavior and surrounding at home). Additionally, two exercises for daily self-guided therapy will be instructed, namely, sit-to-stand and balance performance exercises.
  Arms: intervention group

SUMMARY:
The aim of this monocentric, block-randomized, controlled, open-label, parallel-group study is to assess whether patients presenting to the emergency department (ED) with a fall within the past 7 days would benefit from a physiotherapy intervention, as compared to patients without physiotherapy intervention at the time of ED presentation. Primary objective of this study is to assess "fear of falling" 7 days after ED presentation with versus without a physiotherapy intervention.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥65
* History of falls within the last 7 days
* Presentation to the ED of the University Hospital Basel

Exclusion Criteria:

* Inpatient disposition after ED work-up
* Immobilizing fractures of the lower extremities
* Inability or contraindications to undergo the investigated intervention or follow the study procedures, e.g. due to certain neurological disorders (such as parkinsonism, hemiplegia, severe multiple sclerosis), language problems, psychological disorders, cognitive impairment
* Prior enrolment in this trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Change in short International Falls efficacy scale (sFES-I) | At Day 0 and Day 7 ± 7 days
  Change in the fear of falling between groups at day 7, measured by the short International Falls efficacy scale (sFES-I). It is a 7-item questionnaire where individuals are instructed to score their concern of falling during an activity on a 4 point Likert scale with 1 as not concerned at all and 4 as very concerned. The item scores are summed up to obtain a total, with a higher score indicating a higher fear of falling.

SECONDARY OUTCOMES:
Feasibility of the intervention | At Day 0
  Feasibility of the intervention assessed by a questionnaire filled out by the physiotherapist
Objective functional levels in the intervention group | At Day 0 and Day 7 ± 7 days
  Functional levels measured by SPPB in the intervention group
Satisfaction with ED work-up | Day 7 ± 7 days
  Patients' satisfaction with ED work-up assessed by questionnaire
Change in short International Falls efficacy scale (sFES-I) | At Day 0, Day 7 ± 7 days, Day 21 ± 3 days, Day 42 ± 3 days
  Change in the fear of falling, measured by the short International Falls efficacy scale (sFES-I). It is a 16-item questionnaire where individuals are instructed to score their concern of falling during an activity on a 4 point Likert scale with 1 as not concerned at all and 4 as very concerned. The item scores are summed up to obtain a total, with higher the score, higher being the concern for falling.
Utilization of medical resources | Day 7 ± 7 days, Day 21 ± 3 days, Day 42 ± 3 days
  Comparison of the use of medical resources between both groups (ED visits, GP visits, hospitalization, physiotherapy, imaging; all since inclusion)
Occurence of falls | Day 7 ± 7 days, Day 21 ± 3 days, Day 42 ± 3 days
  Occurence of falls following randomization from patient recollection

CONTACTS AND LOCATIONS:
Overall Officials: Roland Bingisser, Prof. Dr. med., Principal Investigator — Department of Emergency Medicine, University Hospital Basel
Locations (1):
- Department of Emergency Medicine, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Benhamou J, Espejo T, Riedel HB, Dreher-Hummel T, Garcia-Martinez A, Gubler-Gut B, Kirchberger J, Overberg JA, Perrot G, Bingisser R, Nickel CH. On-site physiotherapy in older emergency department patients following a fall: a randomized controlled trial. Eur Geriatr Med. 2025 Feb;16(1):205-217. doi: 10.1007/s41999-024-01091-x. Epub 2024 Nov 16. PMID 39548032